CLINICAL TRIAL: NCT02604992
Title: An Open-Label, Randomized, Single-Dose, Two-Period, Two-Way Crossover Comparative Bioavailability Study of Dronabinol Oral Solution, 4.25 mg to Marinol Capsule, 5 mg in Healthy Volunteers Under Fed Conditions
Brief Title: Comparative Bioavailability of Dronabinol Oral Solution in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: INS004-15-059
Record Dates: First submitted 2015-11-12; First posted 2015-11-16 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: Comparative Bioavailability
MeSH Terms: interventions — Dronabinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1 (A,B,C) (Experimental): With a 7-day washout between periods, participants are randomized to receive Treatment A, Treatment B, and then Treatment C.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Group 2 (B,C,A) (Experimental): With a 7-day washout between periods, participants are randomized to receive Treatment B, Treatment C, and then Treatment A.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Group 3 (C,A,B) (Experimental): With a 7-day washout between periods, participants are randomized to receive Treatment C, Treatment A, and then Treatment B.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Group 4 (C,B,A) (Experimental): With a 7-day washout between periods, participants are randomized to receive Treatment C, Treatment B, and then Treatment A.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Group 5 (A,C,B) (Experimental): With a 7-day washout between periods, participants are randomized to receive Treatment A, Treatment C, and then Treatment B.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Group 6 (B,A,C) (Experimental): With a 7-day washout between periods, participants are randomized to receive Treatment B, Treatment A, and then Treatment C.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C

INTERVENTIONS:
Drug: Treatment A — Dronabinol oral solution, under fed conditions
Drug: Treatment B — Dronabinol oral capsule, under fed conditions
  Other Names: Marinol
Drug: Treatment C — Dronabinol oral capsule, under fasted conditions
  Other Names: Marinol

SUMMARY:
The primary objective of this study is to evaluate the comparative bioavailability of a test product of dronabinol oral solution administered under fed conditions to the reference listed drug (RLD) administered to participants under fed and fasted conditions.

The secondary objective is to compare the onset of detectable dronabinol concentrations between dronabinol oral solution and the RLD.

ELIGIBILITY:
Inclusion Criteria:

* Meets protocol-specified criteria for qualification
* Fully comprehends and signs the informed consent form, understands all study procedures, and can communicate satisfactorily with the Investigator and study coordinator

Exclusion Criteria:

* History or current use of over-the-counter medications, dietary supplements, or drugs outside protocol-specified parameters
* Signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

  1. the safety or well-being of the participant or study staff
  2. the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding)
  3. the analysis of results

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve from time 0 to the last measured concentration | 0 hour (predose), 0.08 (5 min), 0.17 (I0 min), 0.25 (15 min), 0.5 (30 min), 0.75 (45 min), 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 12, and 16 hours postdose.
Area under the curve extrapolated to infinity | 0 hour (predose), 0.08 (5 min), 0.17 (I0 min), 0.25 (15 min), 0.5 (30 min), 0.75 (45 min), 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 12, and 16 hours postdose.
Maximum plasma concentration | 0 hour (predose), 0.08 (5 min), 0.17 (I0 min), 0.25 (15 min), 0.5 (30 min), 0.75 (45 min), 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 12, and 16 hours postdose.
Time to reach maximum plasma concentration | 0 hour (predose), 0.08 (5 min), 0.17 (I0 min), 0.25 (15 min), 0.5 (30 min), 0.75 (45 min), 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 12, and 16 hours postdose.
Elimination rate constant | 0 hour (predose), 0.08 (5 min), 0.17 (I0 min), 0.25 (15 min), 0.5 (30 min), 0.75 (45 min), 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 12, and 16 hours postdose.
The time prior to the first measurable (non-zero) concentration | 0 hour (predose), 0.08 (5 min), 0.17 (I0 min), 0.25 (15 min), 0.5 (30 min), 0.75 (45 min), 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 12, and 16 hours postdose.
Elimination half-life | 0 hour (predose), 0.08 (5 min), 0.17 (I0 min), 0.25 (15 min), 0.5 (30 min), 0.75 (45 min), 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 12, and 16 hours postdose.
Apparent oral clearance | 0 hour (predose), 0.08 (5 min), 0.17 (I0 min), 0.25 (15 min), 0.5 (30 min), 0.75 (45 min), 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 12, and 16 hours postdose.
Volume of distribution | 0 hour (predose), 0.08 (5 min), 0.17 (I0 min), 0.25 (15 min), 0.5 (30 min), 0.75 (45 min), 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 8.0, 12, and 16 hours postdose.

CONTACTS AND LOCATIONS:
Overall Officials: Neha Parikh, Study Director — INSYS Therapeutics Inc
Locations (1):
- Worldwide Clinical Trials Early Phase Services, LLC, San Antonio, Texas, United States